CLINICAL TRIAL: NCT00991874
Title: A Longitudinal Study of Exhaled Nitric Oxide in Children
Acronym: LENOS
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 09/S0801/53
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
Keywords: Nitric oxide; Asthma; Longitudinal studies; Child
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Five percent of children in the UK are prescribed steroid inhalers to control asthma symptoms but there is no test to determine whether the dose of steroids is correct. Too much steroid treatment has potential side effects and too little may lead to asthma attacks. Exhaled nitric oxide (ENO) is a gas present in everyone's breath and may be a useful "meter" for asthma control. In children, ENO can be measured easily and quickly, the results are available immediately to the doctor or nurse and for these reasons ENO is an attractive clinical test.

Pioneering studies have used ENO to help clinicians treat asthmatic adults and children and the results are promising. Breathing tests improved among those where asthma treatment was guided by ENO and asthma symptoms were slightly less frequent. These studies all used a single ENO value to increase or reduce treatment and study authors have suggested there should be a range of ENO values where treatment is neither increased nor reduced; what is not known is what these ENO values may be. Elevated NO is associated with a number of factors other than asthma, including allergy and pollen exposure. What is not known is how factors other than asthma affect ENO measurements over time.

The proposed study will answer two important questions: What values of ENO indicate that steroid treatment should be increased or reduced? And how much does ENO rise and fall normally? The investigators will recruit 200 asthmatic and non-asthmatic children. The investigators will measure ENO on six occasions over a 12-month period. The investigators will measure factors that may affect ENO other than asthma. For the asthmatic children, the investigators will also assess asthma control. The investigators' methodology is based on several years experience with ENO. The investigators' results will allow ENO to be used to monitor asthma.

DETAILED DESCRIPTION:
Our hypotheses are that there will be different ENO values that correlate with loss of/gain in asthma control and that ENO variability is related to environmental exposures including tobacco smoke and pollen. Our research questions are:

1. Do determine what values or % change in ENO correlates with gain and loss of asthma control
2. To determine by how ENO measurements vary within an individual over a 12-month period among children aged 6-16
3. To determine whether ENO measurements vary by the same degree for stable asthmatic, non-asthmatic atopic and non-asthmatic non-atopic children
4. To determine whether variability in ENO correlates with environmental exposures including tobacco smoke, pollen, domestic animals, mould and ambient NO2

Background Asthma is a common chronic condition that affects approximately one million children in the UK and 5% of all children in the UK are prescribed inhaled corticosteroids (ICS) to palliate asthma symptoms. The 2008 British Thoracic Society/Scottish Intercollegiate Guidelines Network guidelines for the management of asthma recommends a step-wise approach to treatment, i.e. treatment is stepped up and down as symptoms relapse and remit. There is no definition of which severity or duration of symptoms should prompt a step-up in treatment. The guideline suggests a "trial and error" approach to stepping down treatment in symptom-free individuals. In the 21st century, the management of asthma remains based on highly subjective clinical decisions and there is a pressing need for a biomarker to guide asthma treatment. "Priorities for respiratory research in the UK" recommends that "Rigorous evaluation is needed of the use of new technologies for diagnostic and monitoring purposes [in asthma], for example exhaled nitric oxide".

A small number of pioneering studies have sought to use ENO to guide asthma treatment, and these have been reviewed recently by the lead applicant. These studies all find ENO-guided treatment is associated with improvements in bronchial hyperresponsiveness, spirometry or ENO. Although all studies found ENO-guided management was associated with improved symptom control, this only achieved significance in one of the four populations studied. The dose of ICS was often considerably higher in individuals where treatment was guided by ENO. One possible reason for the lack of improved symptom control despite increased ICS dose is that all studies used a single cut-off value for ENO to step up or step down ICS treatment; in this situation treatment may be stepped up in an individual with minimal/no symptoms but with a relatively small increase in ENO. Use of separate ENO values for stepping up and stepping down treatment may be more effective, and a recent study has found that changes in paired ENO measurements between -40% and +30% from baseline did not indicate gain or loss of asthma control. Additionally, approximately 10% of individuals with high ENO do not have airway eosinophilia and in this subgroup, who have minor asthma symptoms, ENO does not reduce with ICS treatment. Whilst the present literature suggests that ENO is a promising biomarker for asthma, the findings to date are conflicting and questions remain. In particular, what is still not understood is (i) what values of ENO (or change in ENO) correspond with loss or gain in asthma control? (ii) the variability of ENO over time independent of asthma.

Our study will include rigorous clinical evaluation of participants and will have good statistical power (a weakness of some previous studies). In the proposed study we will take ENO measurements on six occasions over a 12-month period in well-phenotyped asthmatic, non-asthmatic atopic and non-atopic non-asthmatic children. We will describe changes in ENO in the context of asthma control. We will use the results to produce a series of cut-offs for change in ENO measurements in children; analogous to traffic lights there will be a green range (little or no change), amber range (slight increase in ENO), red range (significant increased in ENO). This "traffic light" approach to asthma management is analogous to current asthma management plans where symptoms and peak flows measurements are used. We will also report on changes in ENO in the context of atopy and also environmental exposures including tobacco smoke, pollen, domestic animals, mould and ambient nitrogen dioxide (NO2) levels. In future, and in collaboration with colleagues in primary care, we will use these ranges to design clinical trials where ENO is used to safely monitor asthma. Our data will also be made public and could be used by colleagues to design studies where ENO is used to step-up and step-down corticosteroid treatment in asthmatic children.

c) Experimental design and methods Study design Protocol. Two hundred children aged between 6 and 10 years at enrolment will be recruited from local schools. The initial assessment will take place at hospital and the remaining five will take place at school. The following will be included in the initial phenotyping assessment: height and weight, a standard respiratory questionnaire (ISAAC), Child Asthma Control Test (CACT) for asthmatics, ENO, spirometry, in bronchodilator response and skin prick reactivity. Longitudinal measurements of ENO will thereafter be taken at two monthly intervals. Asthmatic children will complete a CACT at each assessment where changes in asthma medication will also be recorded. The defined primary end point is change in ENO between assessments where asthma control changes. The defined secondary end point will be variability in ENO over 12 months.

Eligibility. Children attending schools in Aberdeen city will be eligible. There is a long tradition of Aberdonian schools and school children participating with asthma studies and we are fortunate to have had the support of Aberdeen City Council, headteachers, class teachers, parents and children over the last 40 years. Our experience is that blanket distribution of letters to parents via class teachers results in relatively poor enrolment rates. We will therefore meet with headteachers and representative of the parent-teachers associations to explain the purpose of the study, gain their approval and include articles in school parent bulletins before approaching the parents and children. Children aged under 6 years will not be included since we have shown that ENO measurements cannot be obtained in the majority of this young age-group. Children who are unable to provide an ENO measurement on the initial assessment will not be included for future assessments. In the event that few children with severe asthma (defined as BTS/SIGN treatment step 3 and 4) are recruited from schools in the first year of the study, we will enrich the cohort with severe asthmatics enrolled from hospital clinics. At the start of the study, written consent will be obtained from parents and verbal assent will be obtained for each assessment from the child.

Categorisation of participants. Children with asthma will be defined as those with affirmative responses to both questions "have you/your child ever had asthma?" and "have you/your child had wheezing or whistling in the chest during the last 12 months?" The number of non-atopic asthmatic children (ie asthma and negative skin prick reactivity) is anticipated to be small; in the final analysis, and only if the number of non-atopic asthmatics is sufficient, we will determine whether the variability for this group differs for the atopic asthmatics. A stable asthmatic will be defined as an asthmatic child where CACT remains ≥19 and treatment does not change over one month.

Questionnaires. At enrolment a validated questionnaire used for the International Study of Allergy and Asthma in Children will be completed. Parents of primary school children (aged≤11 years) will complete the wheezing, rhinitis and eczema modules in the core questionnaire for 6-7 year olds. Children attending secondary schools (aged >12 years) will themselves complete the wheezing, rhinitis and eczema modules in the core questionnaire for 13-14 year olds. Asthmatic children will also complete the CACT. A CACT score of ≥19 will be defined as loss of asthma control. A CACT score of <16 will be used to define good asthma control and has a 79% negative predictive value for physician-defined uncontrolled asthma. Indoor NO2 exposure will be ascertained using questions relating to open gas fires and hobs in the home. Current cat and dog exposure will be defined as an affirmative response to the questions "Do you currently have a cat at home?" and "Do you currently have a dog at home?" Mould exposure will be determined from the response to the "Is there visible damp within the home?" if so which room?" Home will be defined as the residence where the child spends most of the week.

ENO measurements. A portable NO analyser (MINO®, Aerocrine, Sweden) will be used to measure ENO in accordance with manufacturer's recommendations. The same MINO® will be used for each school to eliminate the risk of potential variability for measurements between analysers. Our group has already validated the use of the MINO® for use in children. The child will be asked to inhale through the analyser and the exhale slowly, using the visual and auditory incentives, at 50ml/s for six seconds. In keeping with international guidelines11, we will report the mean ENO from three measurements within 10% or two measurements within 5% of each other; this approach minimises any inherent variability in ENO measurements due to the analyser itself. Measurements will be taken at the same time of day for each child, if possible, and this will eliminate any possible diurnal variability in ENO measurements. Exhaled measurements will not be taken in children who have a concurrent cold since this may affect the ENO result.

Spirometry. Spirometry will be used to phenotype the study participants. A standard portable pneumotachograph (ML3500, MicroLab) will be calibrated and used in accordance with the manufacturer's recommendations, international recommendations will be followed. Each child will complete three forced expiratory manoeuvres, the highest FEV1 and FVC values will be identified, FEV1 and FEV1/FVC ratio will be recorded.

Bronchodilator response. We will measure FEV1 before and 15 minutes after 200 micorg salbutaom (mid/spacer).

Skin Prick Reactivity. The skin prick test will be used to determine reactivity to cat dander, house dust mite, hen's egg, tree pollen, timothy grass, dog dander, cat dander, Aspergillus and Alterneria (allergens provided by ALK, Northampton). Positive (histamine 10mg/ml) and negative controls (0.9% saline) will be used. Atopy will be defined as at least one wheal that measures more than 2mm in longest diameter.

Ambient NO2 concentration. Using the Aberdeen NO2 diffusion tube network we will assess the likely average weekly NO2 exposure for each child in the week in which their measurements were made. This will be supplemented by an assessment of indoor NO2 exposure from questionnaire data.

Pollen exposure. This will be done by looking at the predictable seasonality of pollen production, ie. Tree pollen March/April Grass pollen June/July. Pollen concentrations are not measured in Aberdeen and concentrations in Dundee will be used as a frame of reference and provided at cost (£500) by the National Pollen and Aerobiology Research Unit. The pollen season difference between Aberdeen and Dundee is likely to be very small and insufficient to affect the timing of pollen exposures.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 5-10 years

Exclusion Criteria:

* None

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with and without asthma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Turner, MD, Principal Investigator — University of Aberdeen